CLINICAL TRIAL: NCT03206099
Title: NIAID Centralized Sequencing Protocol
Status: Recruiting | Type: Observational
Sponsor: National Institute of Allergy and Infectious Diseases (NIAID) (NIH)
Collaborators: National Institute of Mental Health (NIMH) (NIH)
Responsible Party: Sponsor
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Other Study IDs: 170122; 17-I-0122
Record Dates: First submitted 2017-06-30; First posted 2017-07-02 (Actual); Last update posted 2026-01-22 (Actual); Status verified 2026-01-20

CONDITIONS: Atopy; Primary Immunodeficiency; Autoimmunity; Autoinflammation
Keywords: Phenotyping; Genetics; Sequencing; Inborn Errors of Immunity; Genomics; Natural History
MeSH Terms: conditions — Primary Immunodeficiency Diseases; Autoimmune Diseases

STUDY DESIGN:
Observational Model: Family Based | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- Biological relatives: Biological relatives of probands, who may or may not also be co-enrolled on the proband's referring protocol.
- Healthy volunteers: Select internal controls
- Probands: Participants with a disease under investigation by another NIAID protocol on which they are enrolled, either at the NIH or CNHS.

SUMMARY:
Background:

Genetic testing called "sequencing" helps researchers look at DNA. Genes are made of DNA and are the instructions for our bodies to function. We all have thousands of genes. DNA variants are differences in genes between two people. We all have lots of variants. Most are harmless and some cause differences like blue or brown eyes. A few variants can cause health problems.

Objective:

To understand the genetics of immune disorders various health conditions, as well as outcomes of clinical genomics and genetic counseling services performed under this protocol.

Eligibility:

Participants in other NIH human subjects research protocols - either at the NIH Clinical Center (CC) or at Children s National Health System (CNHS) - (aged 0-99 years), and, in select cases, their biological relatives

Design:

Researchers will study participant s DNA extracted from blood, saliva, or another tissue sample, including previously collected samples we may have stored at the NIH. Researchers will look at participant s DNA in great detail. We are looking for differences in the DNA sequence or structure between participants and other people.

Participants will receive results that:

* Are important to their health
* Have been confirmed in a clinical lab
* Suggest that they could be at risk for serious disease that may affect your current or future medical management.

Some genetic information we return to participants may be of uncertain importance.

If genetic test results are unrelated to the participant s NIH evaluations, then we will not typically report:

* Normal variants
* Information about progressive, fatal conditions that have no effective treatment
* Carrier status (conditions you don t have but could pass on)

The samples and data will be saved for future research.

Personal data will be kept as private as possible.

If future studies need new information, participants may be contacted.

DETAILED DESCRIPTION:
Investigators at the National Institute of Allergy and Infectious Diseases (NIAID) use next-generation sequencing technologies to help determine genetic contributions to immune diseases. These efforts have increased rates of molecular diagnosis for a subset of NIAID

participants as well as uncovered fundamental insights into the cellular and signaling pathways in host defense and immune regulation.

Despite these successes, analysis and interpretation of genomic data remain a substantial challenge. Simply, researchers do not understand the functional and clinical consequences of most human genetic variation. This is true at NIAID and across the intramural research program. Making progress in this area requires a coordinated, systematic, and transparent approach to clinical genomics research.

This protocol is specific to genetic testing and explicitly aims to both strengthen clinical care and enhance research throughout participating programs at the NIH. Probands will provide biological specimens for genetic testing and will be required to be enrolled on a primary protocol, which will execute the primary clinical and research evaluations. This protocol serves as a vehicle for a

programmatic effort that includes standardized phenotyping, test ordering through the Clinical Research Information System (CRIS), sample collection and isolation, nucleic acid analysis, bioinformatics, clinical interpretation, reporting in CRIS, genetic counseling, and supporting effective use of genomics as a research tool throughout the intramural program. Genetic testing results and data (upon request) will be shared with the research teams for protocols on which a given participant is co-enrolled. Overall, increased process standardization will support data integrity and efficiency while still accommodating the need for investigator flexibility.

ELIGIBILITY:
* PARTICIPANT INCLUSION CRITERIA:
* Must fulfill one of the following criteria:

  * Proband participants: must be individuals under investigation by another NIH protocol on which they are co-enrolled, or are referred from the GDMCC protocol "Defining the Genetic Etiology of Suppurative Lung Disease in Children and Adults" (NCT04702243). Probands may have a disease under investigation or be healthy volunteers
  * Biological relatives: biologically related to a proband participant.
* Aged 0-99 years.
* Participants must be willing to undergo genetic testing.
* Participants must be willing to allow samples to be stored for future research.
* Participants must be willing to have their de-identified genomic data shared, for example in a controlled access databases like the Database of Genotypes and Phenotypes (dbGaP).
* To complete surveys and interviews:

  * Proficient with the English language.
  * Able to provide informed consent.
* Adult healthy volunteers must be able to provide informed consent.

PARTICIPANT EXCLUSION CRITERIA:

Any condition that, in the opinion of the investigator, contraindicates participation in this study is a reason for exclusion.

Ages: 1 Day to 100 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: Probands and their biological relatives (primarily clinical), recruited from NIAID protocols (both at the NIH and CNHS).
Sampling Method: Non-Probability Sample
Enrollment: 20000 (Estimated)
Dates: Start 2017-07-31 (Actual); Primary Completion 2029-12-31 (Estimated); Study Completion 2029-12-31 (Estimated)

PRIMARY OUTCOMES:
Identifying novel genetic defects associated with immune disorders | Upon analysis of genomic data
  Identifying novel genetic defects associated with immune disorders
Identifying novel clinical phenotypes associated with established genetic defects | Upon analysis of genomic data
  Identifying novel clinical phenotypes associated with established genetic defects
Identifying established genetic disorders of the immune system | Upon analysis of genomic data
  Identifying established genetic disorders of the immune system, as well as known genetic disorders outside of the immune system in some cases

SECONDARY OUTCOMES:
Evidence base for how to improve clinical genomic services on this protocol and related programs. | 5.1.1. Enrollment/Baseline Report Comprehension Survey and Semi-Structured Phone Interviews
  Studies of the processes and outcomes of the clinical genomics and genetic counseling services performed under this protocol. These studies will use surveys, interviews, and other social and behavioral research methods to collect data from study participants about their perceptions, experiences, and attitudes related to their condition and participation in this protocol. The goal of these additional studies will be to improve the services provided under protocol 17-I-0122 and to generate an evidence base for other investigators conducting similar studies.

CONTACTS AND LOCATIONS:
Overall Officials: Morgan N Similuk, Principal Investigator — National Institute of Allergy and Infectious Diseases (NIAID)
Locations (2):
- United States (2):
  - Children's National Health System, Washington D.C., District of Columbia
  - National Institutes of Health Clinical Center, Bethesda, Maryland

IPD SHARING:
Plan to Share IPD: Undecided
The PI is on maternity leave and will discuss when they return

REFERENCES:
- [Derived] Zainab R, Kaur S, Lack J, Similuk M, Tandon M, Ghosh R, Seifert BA, Tokita M, Flippo C, Yan J, Walkiewicz M, Chittiboina P, Tatsi C. Genetic evaluation of pediatric pituitary adenomas and USP8-related genotype-phenotype correlations in Cushing's disease. Pituitary. 2025 Aug 14;28(5):92. doi: 10.1007/s11102-025-01557-6. PMID 40813536
- [Derived] Beers BJ, Similuk MN, Ghosh R, Seifert BA, Jamal L, Kamen M, Setzer MR, Jodarski C, Duncan R, Hunt D, Mixer M, Cao W, Bi W, Veltri D, Karlins E, Zhang L, Li Z, Oler AJ, Jevtich K, Yu Y, Hullfish H, Bielekova B, Frischmeyer-Guerrerio P, Dang Do A, Huryn LA, Olivier KN, Su HC, Lyons JJ, Zerbe CS, Rao VK, Keller MD, Freeman AF, Holland SM, Franco LM, Walkiewicz MA, Yan J. Chromosomal microarray analysis supplements exome sequencing to diagnose children with suspected inborn errors of immunity. Front Immunol. 2023 May 5;14:1172004. doi: 10.3389/fimmu.2023.1172004. eCollection 2023. PMID 37215141
- [Derived] Ferre EMN, Yu Y, Oikonomou V, Hilfanova A, Lee CR, Rosen LB, Burbelo PD, Vazquez SE, Anderson MS, Barocha A, Heller T, Soldatos A, Holland SM, Walkiewicz MA, Lionakis MS. Case report: Discovery of a de novo FAM111B pathogenic variant in a patient with an APECED-like clinical phenotype. Front Immunol. 2023 Feb 17;14:1133387. doi: 10.3389/fimmu.2023.1133387. eCollection 2023. PMID 36875114
- [Derived] Similuk MN, Yan J, Ghosh R, Oler AJ, Franco LM, Setzer MR, Kamen M, Jodarski C, DiMaggio T, Davis J, Gore R, Jamal L, Borges A, Gentile N, Niemela J, Lowe C, Jevtich K, Yu Y, Hullfish H, Hsu AP, Hong C, Littel P, Seifert BA, Milner J, Johnston JJ, Cheng X, Li Z, Veltri D, Huang K, Kaladi K, Barnett J, Zhang L, Vlasenko N, Fan Y, Karlins E, Ganakammal SR, Gilmore R, Tran E, Yun A, Mackey J, Yazhuk S, Lack J, Kuram V, Cao W, Huse S, Frank K, Fahle G, Rosenzweig S, Su Y, Hwang S, Bi W, Bennett J, Myles IA, De Ravin SS, Fuss I, Strober W, Bielekova B, Almeida de Jesus A, Goldbach-Mansky R, Williamson P, Kumar K, Dempsy C, Frischmeyer-Guerrerio P, Fisch R, Bolan H, Metcalfe DD, Komarow H, Carter M, Druey KM, Sereti I, Dropulic L, Klion AD, Khoury P, O' Connell EM, Holland-Thomas NC, Brown T, McDermott DH, Murphy PM, Bundy V, Keller MD, Peng C, Kim H, Norman S, Delmonte OM, Kang E, Su HC, Malech H, Freeman A, Zerbe C, Uzel G, Bergerson JRE, Rao VK, Olivier KN, Lyons JJ, Lisco A, Cohen JI, Lionakis MS, Biesecker LG, Xirasagar S, Notarangelo LD, Holland SM, Walkiewicz MA. Clinical exome sequencing of 1000 families with complex immune phenotypes: Toward comprehensive genomic evaluations. J Allergy Clin Immunol. 2022 Oct;150(4):947-954. doi: 10.1016/j.jaci.2022.06.009. Epub 2022 Jun 24. PMID 35753512
- See also: NIH Clinical Center Detailed Web Page — https://clinicalstudies.info.nih.gov/cgi/detail.cgi?A_2017-I-0122.html